CLINICAL TRIAL: NCT00706940
Title: Tear Dynamics After Restasis Treatment in Dry Eye Patients Phase II Clinical Trial and Phase IIb 6-month Follow-up After Discontinuation of Study Treatment
Brief Title: Tear Dynamics After Restasis Treatment in Dry Eye Patients
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jianhua (Jay) Wang, MD, PhD, Associate Professor, University of Miami
Other Study IDs: 20080340
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Dry Eye
Keywords: dry eye; Optical coherence tomography
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observe the changes of tear volume in dry eye patients after Restasis treatment of 3 months and during 6-month follow-up after discontinuation of study treatment.

DETAILED DESCRIPTION:
Using an imaging device name optical coherence tomography to image the tear volume in dry eye patients before and after Restasis treatment.

ELIGIBILITY:
Inclusion Criteria:

The participant will be eligible for entry in the study if s/he:

1. Is at least 18 years old and has full legal capacity to volunteer;
2. Has read and signed the IRB Informed Consent Document;
3. Is willing and able to follow participant instructions;
4. Has clear corneas;
5. Has 20/100 uncorrected visual acuity or better;
6. Has dry eye according to the study definition of DES (study subjects);
7. Has not use Restasis within 3 months.

Exclusion Criteria:

The subjects will ineligible for entry into the study if s/he:

1. Has any systemic disease affecting ocular health except for Sjögren's syndrome;
2. Is using any systemic or topical medications that will affect ocular health except for artificial tears;
3. Has an active ocular disease other than DES, or Sjögren's syndrome
4. Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities;
5. Has limbal or bulbar injection or corneal staining that was clinically significant, which are not due to DES;
6. Has worn rigid gas permeable lenses within 1 year and during the study;
7. Has had surgery or an eye injury within 6 months;
8. Was a soft contact lens wearer within 2 weeks and during the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dry eye patients more than 18 yrs old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Increase in tear volume after the 3-month treatment and returned to baseline during 6-month follow-up after discontinuation of study treatment. | 3 months for treatment and follow-up of 6 months after discontinuation of study treatment.
Tear meniscus volume after treatment | 3 months
  Significant increase in tear meniscus volume was found in patients after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States